CLINICAL TRIAL: NCT00666445
Title: Improved Diagnosis of Alzheimer's Disease Using Magnetoencephalography (MEG) and the Synchronous Neural Interaction™ Test: AD Template Development Study
Brief Title: Improved Diagnosis of Alzheimer's Disease Using the Synchronous Neural Interaction™ Test
Status: Completed | Type: Observational
Sponsor: Orasi Medical, Inc. (Industry)
Collaborators: Noran Neurological Clinic (Unknown); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Todd Verdoorn, Ph.D., Chief Scientific Officer, Orasi Medical, Inc.
Other Study IDs: ADG-08-01
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Diagnosis; Neuronal function; Cognitive Impairment; Magnetoencephalography
MeSH Terms: conditions — Alzheimer Disease; Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients diagnosed with Alzheimer's Disease
- 2: Aged-matched normal controls

SUMMARY:
This study is designed to test the hypothesis that the Synchronous Neural Interaction™ Test is useful for diagnosing Probable Alzheimer's Disease according to standard criteria. Subjects diagnosed with Alzheimer's Disease as well as age-matched normal control subjects will be evaluated for symptoms of Alzheimer's Disease and those meeting inclusion criteria will undergo a brief, non-invasive scan of brain function using a magnetoencephalography (MEG). The scan itself lasts 1 minute while the subject is asked to stare at a dot projected in front of them on a video screen. Orasi Medical believes that patterns of brain activity measured at rest are indicative of Alzheimer's Disease pathology.

The protocol is amended to add a follow-up assessment for previously enrolled and completed subjects who agree to participate in the follow-up assessment approximately 9 - 15 months after initial study enrollment. Subjects who agree to participate in the follow-up assessment will undergo the same standardized tests and MEG scan procedure as completed in the initial study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 90 years of age
2. i. Provide written informed consent for study participation, OR ii. Provide written assent to study participant accompanied by the provision of written informed by the subject's legally authorized representative (LAR); see Section 8. Informed Consent for details of the procedures use to meet these study inclusion criteria
3. Have one of the following clinical diagnoses or conditions:

   * Probable AD according to the NINCDS-ADRDA criteria
   * Possible AD according to the NINCDS-ADRDA criteria
   * Prodromal AD according to criteria described by Dubois & Albert (2004)
   * Normal control subject

Exclusion Criteria:

1. Have a significant non-AD neurological condition including Parkinson's Disease, Vascular Dementia, Lewy Body Dementia or Frontal Temporal Dementia, human immunodeficiency virus, multiple sclerosis, epilepsy, or severe traumatic brain injury.
2. Have dementia due to multiple etiologies (e.g. mixed dementia)
3. Show the presence of prominent disturbances in gait thought to be associated with Parkinsonism.
4. Show prominent changes in personality or social conduct prior to the onset of prominent cognitive dysfunction
5. Have a Modified Hachinski Ischemia Scale score of greater than 4
6. Have a history of primary psychotic disorder (e.g schizophrenia, schizoaffective disorder, delusional disorder) or bipolar disorder
7. Have a lifetime or current history of alcohol or substance abuse/dependence
8. Have had an MRI two weeks prior to completing the MEG scan
9. Have metal braces or pacemaker that may interfere with the MEG scan
10. Are unable to complete the MEG scan procedure

Follow-up Assessment Inclusion Criteria:

Subjects who completed Protocol ADG 08-01 will be contacted and invited to participate in the follow-up assessment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be referred from dementia/Alzheimer's Disease clinical patients at study sites.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for test under investigation to diagnose probable Alzheimer's Disease. | Immediately

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Verdoorn, Ph.D., Principal Investigator — Orasi Medical, Inc.
Locations (3):
- United States (3):
  - Veterans Affairs Medical Center (Brain Science Center), Minneapolis, Minnesota
  - Veterans Affairs Medical Center (Geriatric Research, Education and Clinical Center), Minneapolis, Minnesota
  - Noran Neurology Clinic, Plymouth, Minnesota

REFERENCES:
- [Background] Georgopoulos AP, Karageorgiou E, Leuthold AC, Lewis SM, Lynch JK, Alonso AA, Aslam Z, Carpenter AF, Georgopoulos A, Hemmy LS, Koutlas IG, Langheim FJ, McCarten JR, McPherson SE, Pardo JV, Pardo PJ, Parry GJ, Rottunda SJ, Segal BM, Sponheim SR, Stanwyck JJ, Stephane M, Westermeyer JJ. Synchronous neural interactions assessed by magnetoencephalography: a functional biomarker for brain disorders. J Neural Eng. 2007 Dec;4(4):349-55. doi: 10.1088/1741-2560/4/4/001. Epub 2007 Aug 27. PMID 18057502
- See also: Minnesota Alzheimers Association — http://www.alz.org/mnnd
- See also: Colorado Alzheimers Association — http://www.alz.org/co
- See also: Texas Alzheimers Association — http://www.alz.org/texas